CLINICAL TRIAL: NCT02632864
Title: Feasibility of High Dose PROton Therapy On Unresectable Primary Carcinoma Of Liver: Prospective Phase II Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joon-Hyeok Lee, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-08-004
Record Dates: First submitted 2015-12-07; First posted 2015-12-17 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Liver Neoplasm; Proton Therapy
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton arm (Experimental): Proton beam therapy
  Interventions: Radiation: Proton arm

INTERVENTIONS:
Radiation: Proton arm — Proton beam therapy

SUMMARY:
The standard treatment of unresectable hepatocellular carcinoma (HCC) is transarterial chemoembolization (TACE) or sorafenib. Though the TACE and the agent showed survival benefit in several randomized phase III trials, the benefit was modest.

Recently, radiotherapy (RT), especially conformal and higher dose with the advancement of RT techniques, showed favorable response rate with acceptable local control rate. Based on those promising results, RT was actively applied in HCC who are not indicated with surgery and/or radiofrequency ablation.

Many researchers reported that there is a relationship between RT dose and tumor response rate. RT dose, however, is frequently limited because the complications (like radiation induced liver disease (RILD), radiation induced gastro-duodenal toxicity, etc.) are also closely related with higher exposed RT dose.

Proton beam has characteristic depth-dose distribution contrast to photon, the "Bragg peak". The advantage of this dose distribution could be more highlighted in HCC management, because of the weakness and maintenance importance of liver function itself in HCC patients. In fact, the superior results of proton beam therapy in HCC were constantly reported in several groups as prospectively as well as retrospectively.

In this background, the investigators planned the present study to evaluate the efficacy and safety of proton beam therapy in HCC patients who are not indicated with surgery and/or radiofrequency ablation (RFA).

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma (HCC) patients (Pathologically proven or HCC diagnosed based on American Association for the Study of Liver Diseases (AASLD) guideline)
* Not indicated with surgical resection and/or RFA
* Discussion in tumor board including gastroenterologist, radiologist, radiation oncologist
* Eastern Cooperative Oncology Group performance status 0 to 2 within 1 week before participate
* Adequate bone marrow function (absolute neutrophil count ≥ 1.0 x 109/l, platelet ≥ 30 x 109/l, hemoglobin ≥ 8 g/dl)
* Adequate liver/renal function within 1 week before participate
* Total bilirubin <3.0 mg/dL, Prothrombin time/International normalized ratio <1.7, Albumin≥2.8g/dL, Aspartate aminotransferase/alanine aminotransferase<6 times of upper normal limit Serum creatinine < 1.5 x upper normal limit, glomerular filtration rate > 50 ml/min
* Informed consent
* If viable tumor is single, 1 cm to 10 cm
* Less than 3 nodules
* Child-Pugh class A, B, or early C (score ≤ 10)
* Women of childbearing potential and male participants must agree to practice adequate contraception while on study and for at least 6 months following the last dose of RT

Exclusion Criteria:

* Uncontrolled hepatic encephalopathy
* Previous history of upper abdominal radiotherapy
* Status of pregnancy or breast feeding
* Less than 12 weeks of expected survival
* Uncontrolled ascites
* Combined with disease known as radiosensitive disorder (connective tissue disorder, Ataxia-telangiectasia)
* Hard to maintain stable respiration less than 5 minutes related with respiratory disease
* Combined with uncontrolled severe acute disease other than liver

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
two-year overall survival | two-year after proton beam therapy

SECONDARY OUTCOMES:
1 month objective response rate | 1 month after proton beam therapy
  Modified Response Evaluation Criteria In Solid Tumors (mRECIST) will be used.
3 month objective response rate | 3 months after proton beam therapy
  Modified Response Evaluation Criteria In Solid Tumors (mRECIST) will be used.
6 month objective response rate | 6 months after proton beam therapy
  Modified Response Evaluation Criteria In Solid Tumors (mRECIST) will be used.
1 year progression free survival | one-year after proton beam therapy
  Modified Response Evaluation Criteria In Solid Tumors (mRECIST) will be used.
1 year local progression free survival | one-year after proton beam therapy
  Modified Response Evaluation Criteria In Solid Tumors (mRECIST) will be used.
6 months adverse event | 6 months after proton beam therapy
  Common Terminology Criteria for Adverse Event v4.0 (CTCAE v4.0) will be used.
1 year adverse event | 1 year after proton beam therapy
  Common Terminology Criteria for Adverse Event v4.0 (CTCAE v4.0) will be used.
Baseline Quality of life assessment by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ C-30) | Within 2 week before proton beam therapy started
1 month Quality of life assessment by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ C-30) compared with baseline | 1 month after proton beam therapy
3 month Quality of life assessment by EORTC QLQ C-30 compared with baseline | 3 month after proton beam therapy
6 month Quality of life assessment by EORTC QLQ C-30 compared with baseline | 6 month after proton beam therapy
Baseline Indocyanine green (ICG) | Within 2 week before proton beam therapy started
  ICG Retention rate at 15 minute will be used.
Indocyanine green (ICG) test change compared with baseline | 3 month after proton beam therapy
  ICG Retention rate at 15 minute will be used.
Baseline hepatobiliary phase signal | Within 2 week before proton beam therapy started
  Hepatobiliary phase (20 minute after gadoxetate disodium injection) will be used to evaluate functioning liver volume.
Hepatobiliary phase signal change after proton beam therapy | 3 month after proton beam therapy
  Hepatobiliary phase (20 minute after gadoxetate disodium injection) will be used to evaluate functioning liver volume.

CONTACTS AND LOCATIONS:
Overall Officials: Joon Hyeok Lee, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea